CLINICAL TRIAL: NCT04398446
Title: Coala-T-CBD Study: A Study of the Effect of Hemp-CBD on the Severity and Duration of Chemotherapy-Induced Peripheral Neuropathy in Patients Receiving Neurotoxic Chemotherapy for Non-Metastatic Breast, Uterine, Pancreatic, and Colorectal Cancer and All Stages of Ovarian Cancer
Brief Title: Effect of Hemp-CBD on Patients With CIPN
Acronym: Coala-T-CBD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Main Line Health (Other)
Collaborators: Ananda Hemp, Inc. (Unknown)
Responsible Party: Principal Investigator, Dr. Marisa Weiss, Director, Breast Radiation Oncology, Principal Investigator, Clinical Professor, Main Line Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F/N-R19-3893L
Record Dates: First submitted 2020-04-23; First posted 2020-05-21 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy; Colorectal Cancer Stage II; Colorectal Cancer Stage III; Breast Cancer; Ovarian Cancer; Uterine Cancer; Pancreatic Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Ovarian Neoplasms; Uterine Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hemp-based CBD (Experimental)
  Interventions: Drug: Hemp-based CBD
- Placebo Oral Tablet (Placebo Comparator)
  Interventions: Other: Placebo oral tablet

INTERVENTIONS:
Drug: Hemp-based CBD — 3x Daily dosing for 12 weeks
  Other Names: Ananda Hemp CBD Spectrum Gelcaps
  Arms: Hemp-based CBD
Other: Placebo oral tablet — 3x Daily dosing for 12 weeks
  Arms: Placebo Oral Tablet

SUMMARY:
The purpose of this study is to assess the effect of a hemp-based cannabidiol (CBD) product, Ananda Hemp Spectrum Gelcaps, on the severity and duration of chemotherapy-induced neuropathy (CIPN) among non-metastatic breast, uterine, pancreatic, and colorectal cancer, and all stages of ovarian cancer in patients who received neoadjuvant or adjuvant therapy that included neurotoxic chemotherapeutic agents.

DETAILED DESCRIPTION:
CIPN is a common complication of many effective cytotoxic agents that can negatively impact patients' treatment course and quality of life. The incidence of CIPN in cancer patients receiving multidrug regimens is estimated at 38%, with frequencies approaching 100% with certain known neurotoxic drug classes. Taxanes (e.g., paclitaxel, docetaxel) and platinum-based agents (e.g., oxaliplatin, cisplatin, carboplatin) in particular, are two commonly used chemotherapy classes that are associated with a high incidence of CIPN. Symptoms of chemotherapy-induced peripheral neuropathy include distal extremity numbness, tingling and pain. Chronic, cumulative symptoms can severely impact quality of life and result in dose reductions and/or drug discontinuation in up to 30% of patients.

Consumers use cannabis products for various reasons including pain, stress, anxiety, and insomnia. The neuro-modulatory effects of phytocannabinoids, tetrahydrocannabinol (THC) and cannabidiol (CBD) in particular, have been documented at both the molecular and clinical level. The endocannabinoid system consists of CB1 receptors and CB2 receptors that act as an inhibitory G-protein within the central and peripheral nervous system, respectively. Several animal models have demonstrated the role endocannabinoids play in neuropathic pain development by showing enhanced neuropathic pain with CB1 receptor deletion and reduced manifestations of neuropathic pain with CB2 receptor overexpression. The therapeutic properties of cannabis-based products have also been illustrated in several randomized double-blind trials that have shown significant pain relief versus placebo in the treatment of neuropathy related to diabetes, spinal cord injury, multiple sclerosis, and HIV associated polyneuropathy. Studies specifically looking at the role of CBD in chemotherapy-induced neurotoxicity have shown a neuroprotective effect of CBD in mouse models. Studies have demonstrated that a 14-day dosing regimen of CBD prevented the onset of paclitaxel-induced mechanical and thermal sensitivity.

These intriguing results suggest that cannabinoid agents could potentially reduce the severity and duration of CIPN in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Non-metastatic breast cancer patients who developed CIPN (CTCAE sensory grade 2 or 3, motor grade <2) after receiving taxane-based chemotherapy in pre-operative or post-operative setting.
* Non-metastatic Colorectal cancer patients with high risk stage II and stage III disease who developed CIPN (CTCAE sensory grade 2 or 3, motor grade <2) after receiving oxaliplatin in the adjuvant setting.
* Ovarian cancer patients who developed CIPN (CTCAE sensory grade 2 or 3, motor grade <2) after receiving taxane-containing chemotherapy in the neoadjuvant or adjuvant setting .
* Uterine cancer patients who developed CIPN (CTCAE grade 2 or 3) after receiving taxane-containing chemotherapy in the neoadjuvant or adjuvant setting.
* Non-metastatic pancreatic cancer patients who developed CIPN (CTCAE grade 2 or 3) after receiving taxane-containing chemotherapy in the neoadjuvant or adjuvant setting.

Exclusion Criteria:

* Family history of genetic/familial neuropathy
* Routine use of recreational or medicinal marijuana products (defined as > 4 times per month) or illicit drug use (positive urine drug screen including opioids, cocaine, amphetamines, PCP, LSD)
* Known underlying liver disease (Child-Pugh B or C) or baseline elevation in ALT, AST or total bilirubin ≥1.5 x upper limit of normal
* Patients taking certain medications will be excluded due to potential CBD-drug interaction. CBD may prevent appropriate drug metabolism increasing risk for toxicity. Co-administration of study product and the following medications will be contraindicated and may lead to participant exclusion: clarithromycin, itraconazole, erythromycin, fluconazole, clopidogrel, rifampin, sulfamethoxazole, warfarin, any opioids, warfarin, antiepileptic medications (including carbamazapine, phenytoin, valproic acid, but excepting of gabapentin, clonazepam or diazepam).
* Underlying history of epilepsy/ recurrent seizure disorder or unexplained seizure within past 6 months
* Patients with uncontrolled cardiovascular disease defined by myocardial infarction, stroke or transient ischemic attack, or need for coronary stent placement within past six months.
* Patients with uncontrolled psychiatric illness (who meet DSM-V criteria) or who are at increased risk for suicidality based on baseline Columbia-Suicide Severity Rating Scale.
* Women who are pregnant or breastfeeding or who refuse to practice an effective form of birth control (condoms, diaphragm, birth control pill, IUD)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in pressure/touch sensation during intervention and at follow-up | Every two weeks for twelve weeks during intervention; One month follow-up
  At regular intervals, CIPN will be assessed by Semmes Weinstein Monofilament Examination using Touch-Test Sensory Evaluator Kit to determine pressure sensation.
Change in pain sensation during intervention and at follow-up | Every two weeks for twelve weeks during intervention; One month follow-up
  At regular intervals, CIPN will be assessed by pinprick examination to determine pain sensation.
Change in vibration sensation during intervention and at follow-up | Every two weeks for twelve weeks during intervention; One month follow-up
  At regular intervals, CIPN will be assessed by 128Hz tuning fork vibration test to determine vibration sensation.
Change in quality of life | Every two weeks for twelve weeks during intervention; One month follow-up
  Quality of life will be measured by European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 Questionnaire, a validated 30-item questionnaire to assess treatment impact on quality of life in cancer patients on 4-point scales, where 4 is most severe.
Change in CIPN symptom severity | Every two weeks for twelve weeks during intervention; One month follow-up
  CIPN symptoms will be measured by EORTC QLQ-CIPN20 Questionnaire, validated 20-item questionnaire to assess symptom severity of chemotherapy-induced peripheral neuropathy on 4-point scales, where 4 is most severe.
Change in pain severity | Every two weeks for twelve weeks during intervention; One month follow-up
  Pain severity will be measured by Brief Pain Inventory (BPI) Short Form, validated 9-item questionnaire to assess the severity of pain and the impact of pain on daily functions on 10-point scales, where 10 is most severe.
Change in sleep quality | Every two weeks for twelve weeks during intervention; One month follow-up
  Sleep quality will be measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Questionnaire, validated 8-item questionnaire to assess sleep quality on 5-point scales, where 5 is the most severe.

SECONDARY OUTCOMES:
Receptivity and accrual rate to clinical studies involving cannabis-based substances. | 1 Day
  Receptivity to clinical trials as well as to the use of CBD will be assessed using a questionnaire that will be distributed to all patients at the first encounter. Responses to this questionnaire will provide information regarding in the use of CBD was influencing factor for those who chose to participate or deferring factor for those who decline participation.
Adherence to CBD Products | Daily, 12 weeks
  Adherence will be assessed with a Dosing Diary.
Rate of side effects using medical-grade CBD concentrates | Daily, 12 weeks
  Side effects will be assessed at each encounter clinical evaluation by patient report in a Dosing Diary. All side effects thought to be secondary to CBD will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Marisa Weiss, MD, Principal Investigator — Main Line Health System
Locations (1):
- Lankenau Medical Center, Wynnewood, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee G, Grovey B, Furnish T, Wallace M. Medical Cannabis for Neuropathic Pain. Curr Pain Headache Rep. 2018 Feb 1;22(1):8. doi: 10.1007/s11916-018-0658-8. PMID 29388063
- [Background] Brzezinski K. Chemotherapy-induced polyneuropathy. Part I. Pathophysiology. Contemp Oncol (Pozn). 2012;16(1):72-8. doi: 10.5114/wo.2012.27341. Epub 2012 Feb 29. PMID 23788859
- [Background] Brzezinski K. Chemotherapy-induced peripheral neuropathy. Part II. Prevention. Contemp Oncol (Pozn). 2012;16(3):258-61. doi: 10.5114/wo.2012.29296. Epub 2012 Jul 6. PMID 23788891
- [Background] Saif MW, Reardon J. Management of oxaliplatin-induced peripheral neuropathy. Ther Clin Risk Manag. 2005 Dec;1(4):249-58. PMID 18360567
- [Background] Wang WS, Lin JK, Lin TC, Chen WS, Jiang JK, Wang HS, Chiou TJ, Liu JH, Yen CC, Chen PM. Oral glutamine is effective for preventing oxaliplatin-induced neuropathy in colorectal cancer patients. Oncologist. 2007 Mar;12(3):312-9. doi: 10.1634/theoncologist.12-3-312. PMID 17405895
- [Background] Ward SJ, Ramirez MD, Neelakantan H, Walker EA. Cannabidiol prevents the development of cold and mechanical allodynia in paclitaxel-treated female C57Bl6 mice. Anesth Analg. 2011 Oct;113(4):947-50. doi: 10.1213/ANE.0b013e3182283486. Epub 2011 Jul 7. PMID 21737705